CLINICAL TRIAL: NCT05787002
Title: An Open-label, 2-Period, 2-Sequence Cross-over Study to Assess the Effect of AZD0780 on the Pharmacokinetics of Rosuvastatin in Healthy Participants
Brief Title: A Study to Assess the Effect of AZD0780 on the Pharmacokinetics of Rosuvastatin.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D7960C00002
Record Dates: First submitted 2023-02-23; First posted 2023-03-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dyslipidemia
Keywords: Hypercholesterolemia; elevated Low-density lipoprotein-cholesterol (LDL-C) levels; Drug-drug interaction; Healthy Participants
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Participants will be randomized, in a 1:1 ratio into each of the treatment arms prior to the study commencing. Each participant will receive 2 treatments in total throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence A-B (Experimental): Participants will receive treatments in the following sequence, a single dose of rosuvastatin tablet alone (Treatment A) in period 1, and then a single dose of rosuvastatin tablet + Dose X AZD0780 tablet (Treatment B) in period 2.
  Interventions: Drug: AZD0780; Drug: Rosuvastatin
- Treatment sequence B-A (Experimental): Participants will receive 1 treatment during each study period in the following sequence: a single dose of rosuvastatin tablet + AZD0780 tablet (Treatment B) in period 1 and then a single dose of rosuvastatin tablet alone (Treatment A) in period 2.
  Interventions: Drug: AZD0780; Drug: Rosuvastatin

INTERVENTIONS:
Drug: AZD0780 — AZD0780 will be administered orally as a single dose after an overnight fast of at least 10 hours with approximately 240 mL of water.
Drug: Rosuvastatin — Rosuvastatin will be administered orally as a single dose after an overnight fast of at least 10 hours with approximately 240 mL of water.

SUMMARY:
The purpose of the study is to assess the effect of AZD0780 on the pharmacokinetics of rosuvastatin, and to assess the safety and tolerability of AZD0780 single dose, in healthy participants administered alone and in combination with rosuvastatin.

DETAILED DESCRIPTION:
Eligible participants will be randomized, in a 1:1 ratio into 2 of the treatment arms. Each participant will receive 2 treatments in total throughout the study. The following treatments will be given in randomized order in fasting state:

Treatment A: single dose of rosuvastatin tablet alone

Treatment B: single dose of rosuvastatin tablet + AZD0780 tablet

The study will comprise:

1. A Screening Period of maximum 28 days.
2. Two Treatment Periods up to 3 days
3. A follow-up period of 10 to 12 days after the last administration of the study drug.

Following an overnight fast (minimum 10 hours) participants will receive either of the two treatments and will remain resident in the Clinical Unit until up to 48 hours after dosing of the study drug (up to Day 3).

The total duration of the study will be up to 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female participants (of non-childbearing potential) aged 18 to 60 years, inclusive, with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and must not be lactating
* Participants with BMI between 18 and 30 kg/m^2, inclusive, and weighing between 50 kg and 100 kg, inclusive

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic or renal disease, or any other clinically significant disease or disorder
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, or HIV.
* Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) first vaccination within 30 days prior to randomization and second vaccination within 10 days of screening
* Confirmed Coronavirus disease 2019 (COVID-19) infection at admission, by Polymerase chain reaction (PCR) test
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening
* History or presence of severe allergy/hypersensitivity
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening
* Positive screen for drugs of abuse, alcohol, or cotinine at screening
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of the study drug
* Any clinically significant abnormalities in clinical chemistry, hematology, coagulation, urinalysis results, ECG or vital signs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from 0 to infinity (AUCinf) of Rosuvastatin | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Area under the plasma concentration-curve from 0 to the last quantifiable concentration (AUClast) of Rosuvastatin | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Maximum observed plasma concentration (Cmax) of Rosuvastatin | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Terminal elimination half-life (t½λz) of Rosuvastatin | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Time to reach maximum observed concentration (tmax) of Rosuvastatin | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Apparent total body clearance (CL/F) of Rosuvastatin | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) of Rosuvastatin | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Area under plasma concentration-time curve from 0 to infinity (AUCinf) of AZD0780 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Area under the plasma concentration-curve from 0 to the last quantifiable concentration (AUClast) of AZD0780 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Maximum observed plasma concentration (Cmax) of AZD0780 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Time to reach maximum observed concentration (tmax) of AZD0780 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Terminal elimination half-life (t½λz) of AZD0780 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Apparent total body clearance (CL/F) of AZD0780 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) of AZD0780 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose
  The effect of AZD0780 on the PK of rosuvastatin in healthy participants will be assessed.

SECONDARY OUTCOMES:
Number of participants with Adverse Events | From Screening (≤ 28 days to Day -2) until Follow-up Visit (10 to 12 days post-final dose)
  The safety and tolerability of AZD0780 in combination with rosuvastatin in healthy participants will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis D7960C00002 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7960C00002&attachmentIdentifier=e4eb368c-d073-4e0c-afe4-c99bb2c71978&fileName=PXL_265053_CSR_synopsis_Final_Draft__Redacted_for_Sponsor_01May24.pdf&versionIdentifier=
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://www.astrazenecaclinicaltrials.com/study/D7960C00002/